CLINICAL TRIAL: NCT03930251
Title: Does the Addition of Cognitive Remediation to Coordinated Specialty Care Services Improve Functional Outcome
Brief Title: Cognitive Remediation for Coordinated Specialty Care
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alice Medalia, Professor of Medical Psychology (in Psychiatry) at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7700; 1R34MH118318-01 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-04-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive Remediation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment as Usual (No Intervention): This is the standard coordinated specialty care treatment (without cognitive remediation) that is provided to OnTrackNY clients. This treatment involves psychiatric treatment, employment and educational support, substance abuse treatment, family education and support, CBT-informed individual psychotherapy, and cognitive health support services as needed.
- Clinic-Based Cognitive Remediation (Experimental): Clinic-based cognitive remediation consists of twice weekly group-based and clinician-led sessions.
  Interventions: Behavioral: Clinic-Based Cognitive Remediation
- Partial-Remote Cognitive Remediation (Experimental): Partial-Remote cognitive remediation consists of one weekly group-based, clinician-led session plus independent cognitive practice.
  Interventions: Behavioral: Partial-Remote Cognitive Remediation

INTERVENTIONS:
Behavioral: Clinic-Based Cognitive Remediation — Computer-based exercises targeting impairments in cognitive domains (sensory processing, processing speed, attention, working memory, executive functions) are paired with verbal discussions and group-based activities to strengthen metacognition and bridge newly learned cognitive skills to everyday life. Sessions are led twice weekly by a clinician in small groups.
  Arms: Clinic-Based Cognitive Remediation
Behavioral: Partial-Remote Cognitive Remediation — Computer-based exercises targeting impairments in cognitive domains (sensory processing, processing speed, attention, working memory, executive functions) are paired with verbal discussions and group-based activities to strengthen metacognition and bridge newly learned cognitive skills to everyday life. Sessions are led once weekly by a clinician in small groups and clients gain additional practice by accessing clinician-assigned computer-based exercises independently.
  Arms: Partial-Remote Cognitive Remediation

SUMMARY:
Cognitive remediation (CR) is an evidence-based behavioral skills intervention that targets the cognitive processes underlying functioning in everyday life. It can be used as part of early intervention to reduce cognitive deficits evident at the first episode of psychosis, and has the potential to impact recovery and quality of life. Across Coordinated Specialty Care (CSC) programs, about half of early psychosis participants do not achieve sustained vocational, educational, and/or social recovery; adding CR to CS programs could improve these outcomes. However, models of CR need to be adapted to meet the developmental needs of a younger population and to better fit the CSC model of service delivery. This study of CR implementation will be conducted within the context of OnTrackNY, a network of first-episode psychosis programs that currently offers basic cognitive health evaluation and supportive treatment but not CR.

Intervention content will be designed and refined based on input from multiple stakeholders. The study will assess two delivery approaches to CR, one that delivers CR exclusively "in-clinic/clinician-led" and the other that is "partial-remote/independent" with one in-clinic/clinician-led session per week plus out-of-clinic independent cognitive practice. Nine OnTrackNY programs will be selected and OnTrackNY clinicians will be trained to conduct a cognitive assessment battery and CR. Three programs will be randomly assigned to provide treatment as usual (TAU) and six programs will be randomly assigned to provide both TAU and CR (either "in-clinic/clinician-led" or "partial-remote/independent"). Using de-identified data collected routinely by OnTrackNY for quality improvement/program evaluation, the investigators will examine whether the addition of CR improves functional outcomes for clients with first-episode psychosis, compare the effectiveness of CR delivery methods, and explore whether cognitive improvement is associated with improvement in functioning.

DETAILED DESCRIPTION:
At the time of first-episode, most people with schizophrenia have cognitive impairments that significantly contribute to poor functioning. Early intervention with cognitive remediation (CR), an evidence-based skills intervention that targets cognitive processes, is designed to enhance cognition and functional recovery in people identified as having cognitive health needs. Evidence suggests that provision of CR to those in the early stage of schizophrenia, and in the context of rehabilitation services, results in greater cognitive and functional gains.

OnTrackNY (OTNY) is a New York-based Coordinated Specialty Care (CSC) program that provides early psychosis treatment to young people, between 16 and 30 years of age, who have experienced the onset of non-affective psychosis within two years of beginning treatment. CSC programs provide a significant benefit over usual care, but on average 50% of patients remain disabled after two years. OTNY, like many other CSC programs, provides cognitive health evaluation and supportive treatment but does not routinely offer CR. However, evidence suggests that when cognitive disability is promptly addressed, people show increased self-esteem, engagement in the community and sense of well-being. Therefore, the addition of CR to OTNY may allow treatment to proceed at a faster rate, promote more rapid engagement and mitigate challenges experienced by clients in school or work.

This study aims to:

1. Adapt a 12-week long CR intervention to 2 delivery methods using the input of experts, OnTrackNY mental health clinicians, and clients to improve the acceptability of the intervention content.
2. Examine whether CR can enhance the cognitive and functional outcomes for people with first episode psychosis (FEP) receiving treatment in a CSC program and identified as having cognitive health needs.
3. Compare the effectiveness of "in clinic/clinician-led" and "partial-remote/independent" CR delivery approaches.

This study will occur in phases. In Phase 1, CR content and delivery will be adapted using the input of experts, and training manuals will be created for two intervention approaches. Phase 2 will involve training of mental health clinicians at two OnTrackNY programs to add a formal battery of cognitive assessments and adapted CR. One program will be assigned to deliver CR exclusively "in-clinic" with the aid of a clinician and the other "partial-remote/independent" (one in-clinic session per week with independent cognitive practice). Following quality improvement/program evaluation procedures, the investigators will refine CR based on feedback from providers and clients. Phase 3 will involve nine OnTrackNY programs where clinicians will be trained by researchers to conduct the formal cognitive assessment battery and CR, if applicable. Three programs will be randomly assigned to provide treatment as usual (TAU) and six will be assigned to TAU and CR (either "in-clinic/clinician-led" or "partial-remote/independent").

Referral for cognitive health services will follow routine clinical practice through which clients and their clinicians document cognitive health needs and decide what intervention suits their needs. Clients will be given the option of enrolling in the program's CR intervention. Client characteristics, CR enrollment and outcomes will be made available for quality improvement monitoring and program evaluation in de-identified form. The investigators will examine outcomes for clients identified as having cognitive health needs. To address whether adding CR improves functional outcomes in CSC programs, the investigators will compare measures of community functioning and psychiatric symptom severity across groups. Functional outcome measures will be examined for the time most proximal to CR enrollment and every three months thereafter until study end (range 3-12 months of follow-up depending upon rolling enrollment). Cognition will be measured before and after completion of CR (an average of 3 months) to compare the effectiveness of the two CR delivery approaches and examine whether cognitive improvement is associated with improvement in functioning.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a participating OTNY cognitive remediation program

Exclusion Criteria:

* Not eligible to be enrolled in a participating OTNY cognitive remediation program

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in occupational functioning | At study enrollment and every 3 months through study end, range of time frame 3-12 months
  Change in occupational functioning will be measured with the MIRECC Global Assessment of Functioning (GAF) Occupational Functioning scale. A clinician rates occupational functioning according to the client's primary role (worker, student, or not in labor force/homemaker) on a scale of 1-100 where a higher rating indicates better functioning.
Change in social functioning | At study enrollment and every 3 months through study end, range of time frame 3-12 months
  Change in social functioning will be measured with the MIRECC Global Assessment of Functioning (GAF) Social Functioning scale. A clinician rates the client's average social functioning during the past month on a scale of 1-100 where higher scores indicate better functioning.
Change in psychiatric symptoms | At study enrollment and every 3 months through study end, range of time frame 3-12 months
  Change in symptoms will be measured with the MIRECC Global Assessment of Functioning (GAF) Symptoms scale. A clinician rates psychiatric symptom severity on a scale of 1-100 where a higher rating indicates fewer or less severe psychiatric symptoms.

SECONDARY OUTCOMES:
Change in Average Neurocognition | Before and after completion of cognitive remediation, an average of 3 months
  Neurocognition will be measured with subtests from the Brief Assessment of Cognition in Schizophrenia (BACS) assessing verbal memory, working memory, speed of processing, and executive function and the Continuous Performance Test - Identical Pairs (CPT-IP) for attention/vigilance. All scores will be converted to standardized T scores and averaged together to formulate one measure, Average Neurocognition. The secondary outcome measure will be change in Average Neurocognition from pre to post treatment such that a higher value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Medalia, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (9):
- United States (9):
  - Kings County Hospital Center, Brooklyn, New York
  - Services for the Underserved, Brooklyn, New York
  - Bellevue Hospital Center, New York, New York
  - Washington Heights Community Service, New York, New York
  - Elmhurst Hospital Center, Queens, New York
  - Rochester Psychiatric Center, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - The Institute for Family Health, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
All materials necessary to replicate the adapted cognitive remediation (CR) intervention will be prepared for public sharing. This includes the menu of web-based cognitive exercises employed by CR clinicians and treatment manual for bridging group verbal discussions. De-identified program evaluation data will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories including the National Database for Clinical Trials related to Mental Illness (NDCT). De-identified data will include demographic data, and raw data derived from occupational, social, symptom, and cognitive measures.
Time Frame: A list of all data expected to be collected in the project will be submitted to the NDCT within 6 months of award. Subsequently, descriptive and raw data will be submitted on a semi-annual basis. Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data in NIH repositories may be accessed through the NIH Data Access Committee which reviews data access and submission requests.